CLINICAL TRIAL: NCT01035216
Title: A Phase I Study of GNKG168 Administered by Intravenous Infusion in Patients With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: A Phase I Study of GNKG168 in Patient With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been terminated.
Sponsor: SBI Biotech Co., Ltd. (Industry)
Responsible Party: SBI Biotech Co., Ltd, Theradex (US Representative Agent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G07-10075
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2011-09

CONDITIONS: Leukemia
Keywords: Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL)
MeSH Terms: conditions — Leukemia; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — GNKG168; CPG-oligonucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GNKG168 (Experimental): The starting dose will be 0.25 mg/kg. If the dose is tolerable, subsequent cohorts will be enrolled and treated with 0.5, 0.75, 1.0 and 1.5 mg/kg. If 0.25 mg/kg proves to be intolerable, the dose will be reduced to 0.15 mg/kg.
  Interventions: Drug: GNKG168

INTERVENTIONS:
Drug: GNKG168 — GNKG168 will be administered as a 60 minute IV infusion once daily for 5 days followed by a 9 day rest period.
  Other Names: CpG ODN

SUMMARY:
This is an open-label, dose escalation study designed to characterize the safety, tolerability, efficacy, and pharmacokinetics of GNKG168 in patients with B-CLL that has relapsed or is refractory to all prior standard therapy, or for which no standard therapy exists.

DETAILED DESCRIPTION:
This is an open-label, dose escalation study designed to characterize the safety, tolerability, efficacy, and pharmacokinetics of GNKG168 in patients with B-CLL that has relapsed or is refractory to all prior standard therapy, or for which no standard therapy exists.

As secondary objectives, baseline TLR-9 intracellular staining of B-CLL cells, and in vitro assays to assess the potential of B-CLL cells to undergo apoptosis in conjunction with GNKG168 therapy will be examined. Baseline characteristics of B-CLL will be examined including interphase genetics, FISH CLL, IgVH mutational status, expression of ZAP70, β2-microglobulin and the expression of the prognostic marker CD38 in peripheral blood cells (at baseline and during treatment) and baseline immune SNPs (FcγRIIIa, FcγRIIa, TNF-α, IFN-γ, CD40 and others). As pharmacodynamics parameters, the expression of B-cell and T-cell activation markers (including IL-21 receptor upregulation), NK cell markers, and cytokines will be investigated.

This clinical trial will also assess the ability of B CLL patients treated with GNKG168 to elicit anti pneumococcal antibodies in response to adjuvant vaccination with the Prevnar™ vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have cytologically confirmed B-cell chronic lymphocytic leukemia (B-CLL) that has relapsed or been refractory to all prior standard therapy, or for which no standard therapy exists, or patients who refuse available therapy.
2. Patients' B-CLL must be staged according to either the Rai or Binet systems23 (see Appendix III) and assessed for chromosomal abnormalities, unmutated IgVH status, and expression of ZAP70, and expression of CD38 (see Section 7.2 Pre-treatment).
3. Patients must have recovered from all acute adverse effects of prior therapies to grade 1, excluding alopecia.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Patients must be ≤ to 18 years of age.
6. Patients must have normal organ function as defined by:

   total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT)≤ 2.5 x ULN serum creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal. The creatinine clearance in male patients may be calculated using the Cockcroft-Gault formula: CrCl (mL/min) = [(140 - age) x weight (kg)]/ 72 x Cr (mg/dL). Note: in female patients, this calculation must be multiplied by a factor of 0.85.
7. Patients must have serum sodium levels ≥ 135 mmol/L and serum chloride levels ≥ 98 mmol/L.
8. Male patients must have a QTc interval of < 450 msec and female patients must have a QTc interval of < 470 msec.
9. Patients must be able to understand and willing to sign a written informed consent document.
10. Patients must be at least 2 weeks from prior chemotherapy, radiation therapy, major surgery, or other investigational anticancer therapy. Patients may receive steroids to control the secondary effects of CLL such as autoimmune cytopenia or painful lymph nodes if this is considered by the treating physician to be in the best interest of the patient.
11. Women of childbearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study. Male and female patients must use acceptable contraceptive methods during the entire study period and for 1 month after the end of study or after being discontinued from the study.

Exclusion Criteria:

1. Patients who are currently receiving chemotherapy, radiotherapy, biological therapy, or any other investigational therapy.
2. Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse effects due to agents administered more than 4 weeks earlier.
3. Patients with uncontrolled known leukemic meningitis, because of their poor prognosis and likelihood of developing progressive neurologic dysfunction which would confound evaluation of neurologic and other adverse events.
4. Patients with a history of sensitivity or allergy attributed to compounds of similar chemical composition to GNKG168 or to the Prevnar™ vaccine.
5. Patients with concurrent serious infections (i.e., requiring an intravenous antibiotic).
6. Patients with active malignancy (excepting non-melanomatous skin cancers) which may limit survival to less than 2 years.
7. Patients with pre-existing autoimmune diseases (i.e. systemic lupus erythematosis, rheumatoid arthritis, Crohn's disease or ulcerative colitis, primary sclerosing cholangitis, thyroiditis, scleroderma, etc.) are not eligible.
8. Women who are pregnant or are of childbearing potential and not using methods to avoid pregnancy, and women who are breastfeeding.
9. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patients with significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within six months of study entry, uncontrolled dysrhythmias or poorly controlled angina.
11. Patients with known positive status for HIV or active hepatitis B or hepatitis C.
12. Patients with any medical condition which in the opinion of the Investigator places them at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicity (DLT) and recommended phase 2 dose

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Univ. of San Diego: Moores UCSD Cancer Center, La Jolla, California
  - University of Minnesota, Minneapolis, Minnesota
  - North Shore University Hospital, New Hyde Park, New York
  - Cornell University, New York, New York
  - Oregon Health & Sciences University, Portland, Oregon